CLINICAL TRIAL: NCT07027436
Title: Radiation Therapy Followed by Durvalumab (MEDI4736) and Tremelimumab And Surgery Versus Radiation Therapy Followed by Surgery for Resectable Hepatocellular Carcinoma. A Randomized Window of Opportunity Trial (DARTS)
Brief Title: Radiation Therapy Followed by Durvalumab (MEDI4736) and Tremelimumab And Surgery Versus Radiation Therapy Followed by Surgery for Resectable Hepatocellular Carcinoma.
Acronym: DARTS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Pablo Serrano, Local principal Investigator, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DARTS ESR-23-22174; ESR-23-22174 (Other: McMaster University)
Record Dates: First submitted 2025-06-03; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Durvalumab/tremelimumab, SBRT, radiation, HCC; WOO, Window of Opportunity
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Drug Therapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT and Chemotherapy (Experimental): Study participants randomized to treatment Group 1, will receive SBRT prior to surgery on Day 1, and receive one infusion of Durvalumab (1500mg IV) / Tremelimumab 300mg IV) on Day 15.
  Interventions: Drug: Chemotherapy/Radiation
- SBRT alone (No Intervention): The patients receive radiation only without chemotherapy SBRT prior to the surgery.

INTERVENTIONS:
Drug: Chemotherapy/Radiation — Combination of radiation and chemotherapy
  Other Names: Group 1
  Arms: SBRT and Chemotherapy

SUMMARY:
The objectives of this study is to estimate the biological activity of combination chemotherapy and radiation versus radiation alone in patients with Hepato Cellular Carcinoma (HCC).

The study hypothesizes is that combination chemotherapy and radiation is superior to radiation alone in inducing a biological response. The study hypothesizes that combination chemotherapy and radiation is superior to radiation alone in inducing a biological response. A biological response, or change in the tumor microenvironment (TME), is defined by reduced infiltration of intra-tumoral regulatory T cells (Tregs), a decrease in tumour-associated macrophages (TAMs) of the M2 phenotype, and an increase in immune cells such as effector CD8+ T-cells. An increased rate of biological response is therefore expected in participants receiving the combination of Durvalumab, Tremelimumab, and stereotactic body radiation therapy (SBRT), compared to those receiving SBRT alone. Additionally, biological response is hypothesized to correlate with pathological response.

The study has been conducted within a WOO window of opportunity randomized clinical trial in order to obtain data in the quickest and safest manner. Patients undergoing surgery are very healthy by definition and will be able to tolerate treatment without any major complications, leading to adequate tissue samples before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically or biopsy proven solitary HCC without biliary invasion or metastases, Liver Imaging Reporting and Data Systems (LI- RADS) 4 or 5 only. Participants with satellite tumour nodules are eligible. Satellitosis or a satellite nodule is defined as a tumour (LI-RADS 4 or 5 only) less than or equal to 2 cm and located less than or equal to 2 cm from the main tumour.

Tumour less than 12 cm in maximum size on CT or MRI.

Planned surgical resection of HCC with a life expectancy of at least 12 weeks

Age >18 years at time of study entry.

Child-Pugh Class A within 14 days prior to study enrollment

Eastern Cooperative Oncology Group (ECOG) of 0 or 1 (see Appendix 3)

Body weight >30 kg at time of study enrollment

Adequate normal organ and marrow function as defined below:

Haemoglobin ≥9.0 g/dL

Absolute neutrophil count (ANC ≥1.0 × 109 /L)

Platelet count ≥75 × 109/L

Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN).

AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal

Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine clearance CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

Males:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age)72 x serum creatinine (mg/dL)

Females:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)

Patient is capable and willing to provide signed informed consent.

Exclusion Criteria:

* Previous therapy for HCC, including systemic therapy, surgery, radiation therapy, ablation or embolization.

Participation in another clinical study with an investigational product during the last 4 weeks or concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.

Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.

Previous radiation therapy or surgery within 4 weeks of the randomization.

Previous allogenic organ transplantation

Previous anti-PD-1, anti-PD-L1 or anti-CTLA-4 therapy

Previous receipt of durvalumab and / or tremelimumab or allergy to it

Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy except for alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.

Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.

Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

Patients with vitiligo or alopecia

Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement

Any chronic skin condition that does not require systemic therapy

Patients without active disease in the last 5 years may be included but only after consultation with the study physician

Patients with celiac disease controlled by diet alone

History of active primary immunodeficiency

Conditions that would preclude administration of durvalumab and / or tremelimumab

Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent

Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Patients with a past or resolved HBV infection (defined as the presence of antiHBc and absence of HBsAg) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.

b.1. Patients co-infected with HBV and HCV or co-infected with HBV and HDV, namely: HBV positive (presence of HBsAg and/or anti HBcAb with detectable HBV DNA); and

b.2. HCV positive (presence of anti-HCV antibodies); or

b.3. HDV positive (presence of anti-HDV antibodies)

b.4. Patients with HBV infection, characterized by positive HBsAg and/or anti-HBcAb with undetectable HBV DNA (< 10 IU/ml or under the limit of detection per local lab standard) do not require antiviral therapy prior to enrollment. These patients will be tested once for HBV DNA levels; if HBV DNA is detected (≥ 10 IU/ml or above the limit of detection per local lab standard), antiviral therapy must be initiated, continued for the study duration and for 6 months after the last dose of IP.

Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) which is not well controlled or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).

c.1. All of the following criteria are required to define an HIV infection that is well controlled: undetectable viral RNA load for 3 months, CD4+ count of >200 no history of AIDS-defining opportunistic infection within the past 12 months, and stable for at least 3 months on the same anti-HIV medications.

History of another primary malignancy, except for

Malignancy treated with curative intent and with no known active disease ≥2 years before randomization and of low potential risk for recurrence

Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease

Adequately treated carcinoma in situ without evidence of disease

Current or prior use of immunosuppressive medication within 14 days before enrollment. The following are exceptions to this criterion:

Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)

Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent

Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)

Receipt of live attenuated vaccine within 30 days prior to enrollment. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 90 days after the last dose of IP.

Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab and tremelimumab combination therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-07 (Estimated); Primary Completion 2027-10-12 (Estimated); Study Completion 2028-10-10 (Estimated)

PRIMARY OUTCOMES:
Intratumoral immune cells (regulatory T lymphocytes or Tregs). | Baseline and immediately after the intervention
  This will be measured pre and post treatment through proteomic analysis with digital spatial profiling (DSP) technology. This will determine with high resolution the area of infiltration (tumour versus stroma), to assess the relative immune status of the tumor (i.e., hot or cold). The primary endpoint is the percentage change in Tregs in the TME. The percentage change in Tregs is defined as the: (number of Tregs at surgery) / (number of Tregs at baseline) *100%.

SECONDARY OUTCOMES:
Intratumoural immune cells including M2-TAMs measured similarly to the primary outcome measure. | Baseline and immediately after the intervention
  measured similarly to the primary outcome measure.
Intratumoural immune cells | Baseline and immediately after the intervention
  Intratumoural immune cells (such as B cells, CD8+ T cells)
TMB | Baseline and immediately after the intervention
  which will be defined as the number of somatic nonsynonymous mutations or variants present in the coding region expressed as mutations per megabase (muts/Mb) of sequence. TMB will be measured using DNA/RNA seq, which will be analysed in the specimen pre- treatment. RNA seq will be analysed post treatment using ThermoFisher's Oncomine Comprehensive Assay Plus Assay (DNA-seq) and ThermoFisher's Ion AmpliSeqTM Transcriptome Human Gene Expression Kit (RNA-seq).
PD-L1 expression | Baseline and immediately after the intervention
  PD-L1 expression before and after treatment will be performed using immunohistochemistry in the specimen
The percent change in peripheral blood immune repertoire. | Baseline and immediately after the intervention
  TCR-sequencing using ThermoFisher's Oncomine TCR Beta-LR Assay: changes in the immune repertoire produced by therapy will be analysed in peripheral blood using DNA from the buffy coat at baseline and post treatment. Relevant T cell clonotypes will be identified through TCR analysis of the resected tumour.

OTHER OUTCOMES:
Exploratory outcome | Baseline and immediately after the intervention
  Pathologic response

CONTACTS AND LOCATIONS:
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No